CLINICAL TRIAL: NCT00611572
Title: Contribution of Gabaergic and Glutamatergic Mechanisms to Cognitive Dysfunction
Brief Title: GABA-glutamate Interactions and Psychosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Alliance for Research on Schizophrenia and Depression (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Other
Other Study IDs: 0508000517
Record Dates: First submitted 2008-01-29; First posted 2008-02-11 (Estimated); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Cognitive Dysfunction
Keywords: GABA; glutamate; NMDA; P300; MMN
MeSH Terms: conditions — Cognitive Dysfunction | interventions — iomazenil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Active iomazenil and ketamine
  Interventions: Drug: iomazenil
- 2 (Placebo Comparator): placebo iomazenil and ketamine
  Interventions: Drug: iomazenil

INTERVENTIONS:
Drug: iomazenil — Given as IV infusion
  Arms: 1
Drug: iomazenil — saline IV infusion
  Arms: 2

SUMMARY:
This study investigates the interactions between NMDA (N-Methyl-D-aspartic acid) antagonism and GABA (gamma-aminobutyric acid) system as it relates to cognitive function assessed by ERPs (event-related potentials) in healthy volunteers.

ELIGIBILITY:
Inclusion criteria:

* Ages of 21-45 years from all ethnic backgrounds.
* Male or female.
* Written informed consent.

Exclusion criteria:

* DSM-IV diagnosis for a psychotic, depressive or anxiety disorder.
* A history of significant medical/neurological disease such as cardiac, thyroid, renal, hepatic abnormality, seizure disorder. Unstable medical condition based on EKG, vital signs, physical examination and laboratory work-up (CBC with differential, SMA-7, LFTs, TFTs, UA, Utox).
* History of abnormal EEG.
* History of severe allergies or multiple adverse drug reactions.
* Any medication that could interfere with either the safety of the study and/or the outcome measures.
* Any other conditions which in the opinion of the investigator would preclude participation in the study.
* History of major psychiatric disorder in first degree relatives.
* Current substance abuse/dependency determined by urine toxicology.
* Treatment with medications with CNS effects.
* Treatment with benzodiazepines within one week prior to testing.
* Current treatment with medications with psychotropic effects.
* Education < 10th grade.
* IQ < 70, MR.
* Non-English speaking.

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2007-01; Primary Completion 2018-10-02 (Actual); Study Completion 2018-10-02 (Actual)

PRIMARY OUTCOMES:
P300 as an ERP measure | prospective

SECONDARY OUTCOMES:
MMN (Mismatch Negativity) | prospective

CONTACTS AND LOCATIONS:
Overall Officials: Mohini Ranganathan, M.D., Principal Investigator — Yale School of Medicine, Associate Professor
Locations (1):
- VHA Connecticut, West Haven, Connecticut, United States